CLINICAL TRIAL: NCT01233869
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study Of The Safety, Clinical Activity And Pharmacokinetics Of Bosutinib (PF-05208763) Versus Placebo In Subjects With Autosomal Dominant Polycystic Kidney Disease (ADPKD)
Brief Title: Bosutinib For Autosomal Dominant Polycystic Kidney Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B1871019; 3160A7-2211 (Other: Alias Study Number); 2010-023017-65 (EudraCT Number)
Record Dates: First submitted 2010-10-28; First posted 2010-11-03 (Estimated); Results first posted 2015-10-28 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-02

CONDITIONS: Polycystic Kidney, Autosomal Dominant
Keywords: Bosutinib; Autosomal Dominant Polycystic Kidney Disease
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant | interventions — bosutinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort A (Experimental)
  Interventions: Drug: Bosutinib
- Cohort B (Experimental)
  Interventions: Drug: Bosutinib
- Cohort C (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bosutinib — Once daily oral dose of 200 mg of bosutinib
  Arms: Cohort A
Drug: Bosutinib — Once daily oral dose of 400 mg of bosutinib transitioned to 200 mg/day
  Arms: Cohort B
Drug: Placebo — Once daily oral dose of placebo
  Arms: Cohort C

SUMMARY:
This purpose of this study is to determine if bosutinib reduces the rate of kidney enlargement in subjects with autosomal dominant polycystic kidney disease (ADPKD) entering the study with a total kidney volume greater than or equal to 750 cc and eGFR greater than or equal to 60 mL/min/1.73m2.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18 to 50 years old at the time of consent.
* Documented diagnosis of ADPKD (PKD-1 or PKD-2 genotypes allowed).
* Total kidney volume ≥ 750 cc, as measured by centrally evaluated MRI.

Exclusion Criteria:

* eGFR < 60 mL/min/1.73m2.
* Uncontrolled hypertension (defined as systolic blood pressure ≥140 or diastolic blood pressure ≥90 mm Hg).
* Any previous exposure to the bosutinib test article or receipt of other polycystic kidney disease (PKD) therapies.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 172 (Actual)
Dates: Start 2010-12; Primary Completion 2014-07 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (67):
- United States (20):
  - Southwest Kidney Institute, PLC, Phoenix, Arizona
  - Southwest Clinical Research Institute, LLC, Tempe, Arizona
  - Southwest Kidney Institute, PLC, Tempe, Arizona
  - Capital Nephrology Clinical Research, Sacramento, California
  - Boise Kidney & Hypertension Institute, PLLC, Caldwell, Idaho
  - Boise Kidney & Hypertension Institute, PLLC, Meridian, Idaho
  - Renal Associates of Baton Rouge, Baton Rouge, Louisiana
  - Tufts Medical Center, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Washington University, St Louis, Missouri
  - New York University - HHC CTSI Clinical Research Center, New York, New York
  - Doylestown Hospital MRI, Doylestown, Pennsylvania
  - Doylestown Hospital, Doylestown, Pennsylvania
  - Nephrology/Hypertension Specialists, Doylestown, Pennsylvania
  - Renal Associates, PA, San Antonio, Texas
  - San Antonio Kidney Disease Center Physicians Group, P.L.L.C., San Antonio, Texas
  - University of Virginia Health System - Nephrology, Charlottesville, Virginia
  - University of Virginia Health System, Charlottesville, Virginia
  - The Polyclinic, Seattle, Washington
  - Renal Remission and Hypertension Clinic, Silverdale, Washington
- Monash Medical Centre, Clayton, Victoria, Australia
- Canada (2):
  - Toronto General Hospital, Toronto, Ontario
  - Hopital du Sacre-Coeur de Montreal, Montreal, Quebec
- Czechia (6):
  - Klinika gerontologicka a metabolicka, Hradec Králové
  - Krajska nemocnice Liberec, Liberec
  - Nemocnice Nove Mesto na Morave, Nové Město na Moravě
  - Fakultni poliklinika VFN, Prague
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Pharmaceutical Research Associates CZ, s.r.o., Prague
- Hungary (3):
  - PRA Magyarorszag Kft. Klinikai Farmakologiai Vizsgalohely, Budapest
  - Fovarosi Onkormanyzat Szent Imre Korhaz BSZMI Klinikai Farmakologiai Reszlege, Budapest
  - Szegedi Tudomanyegyetem, AOK, Szent-Gyorgyi Albert Klinikai Kozpont I.sz.Belgyogyaszati Klinika, Szeged
- Italy (2):
  - Istituti Ospitalieri di Cremona, Cremona
  - A.O. Universitaria Ospedali Riuniti di Foggia, Foggia
- Vilnius University Hospital Santariskiu Clinic, Public Institution, Centre of Nephrology, Vilnius, Lithuania
- Spitalul Clinic Republican, Chisinau, Moldova
- Poland (11):
  - Zaklad Diagnostyki Chorob Serca, II Katedra Kardiologii, Gdansk
  - Klinika Nefrologii, Transplantologii i Chorob Wewnetrznych, Gdansk
  - Specjalistyczny Szpital Zachodni im. Jana Pawla II w Grodzisku Mazowieckim, Grodzisk Mazowiecki
  - Krakowskie Centrum Medyczne NZOZ, Krakow
  - Klinika Nefrologii, Hipertensjologii i Chorob Wewnetrznych Katedry Chorob Wewnetrznych UWM, Olsztyn
  - Pracownia Echokardiografii, Oddzial Kardiologii, Olsztyn
  - Centrum Medyczne Aesculap, Radom
  - Klinika Kardiologii, Szczecin
  - Klinika Nefrologii, Transplantologii i Chorob Wewnetrznych, Szczecin
  - Szpital Powiatowy w Wolominie, Wołomin
  - SPZOZ Akademicki Szpital Kliniczny im. J. Mikulicza - Radeckiego, Wroclaw
- Romania (4):
  - Spitalul Clinic Municipal Dr. Gavril Curteanu Oradea, Oradea, Jud. Bihor
  - Spitalul Clinic Dr. C. I. Parhon Iasi, Iași, Jud. Iasi
  - Institutul Clinic Fundeni, Centrul de Medicina Interna-Nefrologie, Bucharest
  - SPITALUL CLINIC JUDETEAN DE URGENTA TIMISOARA ,Clinica de Nefrologie, Timișoara
- Slovakia (2):
  - Univerzitna nemocnica Bratislava, Limbova 5, Bratislava Region
  - SUMMIT CLINICAL RESEARCH, s.r.o., Oddelenie internej mediciny a klinickej farmakologie, Bratislava
- South Korea (3):
  - Seoul National University Hospital, Department of Internal Medicine, Seoul
  - Samsung Medical Center/Division of Nephrology, Seoul
  - Eulji General Hospital, Seoul
- Spain (2):
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Clinic I Provincial de Barcelona, Barcelona
- Sweden (3):
  - Sahlgrenska Universitetssjukhuset, Njurmedicin, Gothenburg
  - Karolinska Universitetssjukhuset Huddinge, Stockholm
  - Karolinska Universitetssjukhuset Solna, Stockholm
- Universitaetsspital Zuerich, Zurich, Switzerland
- Turkey (Türkiye) (2):
  - Istanbul University, Istanbul Tip Fakultesi, Istanbul, Capa
  - Dokuz Eylul Universitesi Hastanesi Ic Hastaliklari Anabilim Dali, Izmir, Inciralti/ Narlidere
- United Kingdom (3):
  - Morriston Hospital, Swansea, Wales
  - BHF Glasgow Cardiovascular Research Centre, University of Glasgow, Glasgow
  - Renal and Urology Directorate, Leicester General Hospital, Leicester

REFERENCES:
- [Derived] St Pierre K, Cashmore BA, Bolignano D, Zoccali C, Ruospo M, Craig JC, Strippoli GF, Mallett AJ, Green SC, Tunnicliffe DJ. Interventions for preventing the progression of autosomal dominant polycystic kidney disease. Cochrane Database Syst Rev. 2024 Oct 2;10(10):CD010294. doi: 10.1002/14651858.CD010294.pub3. PMID 39356039
- [Derived] Tesar V, Ciechanowski K, Pei Y, Barash I, Shannon M, Li R, Williams JH, Levisetti M, Arkin S, Serra A. Bosutinib versus Placebo for Autosomal Dominant Polycystic Kidney Disease. J Am Soc Nephrol. 2017 Nov;28(11):3404-3413. doi: 10.1681/ASN.2016111232. Epub 2017 Aug 24. PMID 28838955
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1871019&StudyName=Bosutinib%20For%20Autosomal%20Dominant%20Polycystic%20Kidney%20Disease

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 172 participants were enrolled in this study, of which 169 received at least 1 dose of study treatment.
Groups:
- Bosutinib 200 mg/Day: Participants received bosutinib 200 mg tablet orally once daily (QD) in the morning with food for 24 months in the Initial Treatment Period (ITP). After a 30-day washout period, participants who entered the Extended Treatment Period (ETP) continued to receive bosutinib 200 mg orally QD for up to 46 months.
- Bosutinib 400 mg/Day: Participants received bosutinib 400 mg tablet orally QD in the morning with food for 24 months in the ITP. All participants were dose-reduced during the ITP based on a protocol amendment. Those who remained active in the study at the time of the amendment are represented in the bosutinib 400/200 mg/day group.
- Bosutinib 400/200 mg/Day: Participants received bosutinib 400 mg and were dose-reduced to 200 mg tablet (based on protocol amendment) orally QD in the morning with food for 24 months in the ITP. After a 30-day washout period, participants who entered the ETP continued to receive bosutinib 200 mg orally QD for up to 46 months.
- Placebo: Participants received placebo tablet orally QD in the morning with food for 24 months in the ITP. After a 30-day washout period, participants who entered the ETP continued to receive placebo matched bosutinib QD for up to 46 months.
Period: Initial Treatment Period (24 Months)
Arm/Group | Bosutinib 200 mg/Day | Bosutinib 400 mg/Day | Bosutinib 400/200 mg/Day | Placebo
Started | 58 | 31 | 24 | 56
Completed | 34 | 3 | 22 | 34
Not Completed | 24 | 28 | 2 | 22
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Adverse Event | 9 | 17 | 0 | 3
Not completed — Not Related to Study Drug | 14 | 11 | 2 | 19
Period: Washout Period 30 Days
Arm/Group | Bosutinib 200 mg/Day | Bosutinib 400 mg/Day | Bosutinib 400/200 mg/Day | Placebo
Started | 34 | 3 | 22 | 34
Completed | 34 | 3 | 22 | 34
Not Completed | 0 | 0 | 0 | 0
Period: Extended Treatment Period (46 Months)
Arm/Group | Bosutinib 200 mg/Day | Bosutinib 400 mg/Day | Bosutinib 400/200 mg/Day | Placebo
Started | 34 | 3 | 22 | 34
Completed | 20 | 0 | 17 | 18
Not Completed | 14 | 3 | 5 | 16
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 10 | 3 | 5 | 11
Not completed — Other | 3 | 0 | 0 | 3
Not completed — Adverse Event | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The safety population included all participants who received at least 1 dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Bosutinib 200 mg/Day | Bosutinib 400 mg/Day | Bosutinib 400/200 mg/Day | Placebo | Total
Number analyzed (Participants) | 58 | 31 | 24 | 56 | 169
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.9 (8.0) | 41.3 (4.9) | 36.4 (7.8) | 38.5 (7.4) | 38.5 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 14 | 15 | 35 | 92
  Male | 30 | 17 | 9 | 21 | 77

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (CFB) in Total Kidney Volume (TKV) at Month 25
Description: TKV was measured by centrally evaluated Magnetic Resonance Imaging (MRI).
Time Frame: Baseline and Month 25 (end of Initial Treatment Period Visit [ITPV])
Population: The modified intent-to-treat (mITT) population included all participants who were randomized and received at least 2-weeks' worth of treatment and have at least 1 follow-up MRI assessment that was preceded by a 1-month washout of the study drug; n=the number of participants analyzed at that time point in the respective arms.
Measure: Mean (Standard Deviation); unit: centimeter cube (cm^3)
Arm/Group | Bosutinib 200 mg/Day | Bosutinib 400 mg/Day | Bosutinib 400/200 mg/Day | Placebo
Number analyzed (Participants) | 27 | 6 | 21 | 33
centimeter cube (cm^3)
  Baseline (n=27,6,21,33) | 1686.38 (944.30) | 1418.96 (629.34) | 1487.48 (531.96) | 1670.33 (640.69)
  CFB at Month 25 (n=23,3,20,30) | 85.05 (231.09) | 102.45 (257.30) | -6.18 (119.79) | 175.36 (191.43)
Statistical Analysis 1: Comparison: Bosutinib 200 mg/Day vs Bosutinib 400 mg/Day vs Bosutinib 400/200 mg/Day vs Placebo; Statistical Analysis 1 is comparison of annualized rate of kidney enlargement: placebo versus pooled bosutinib; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Median Difference (Final Values) = 3.86, 95% CI 2-sided [2.02 to 5.74]
Statistical Analysis 2: Comparison: Bosutinib 200 mg/Day vs Bosutinib 400/200 mg/Day; Statistical Analysis 2 is comparison of annualized rate of kidney enlargement: bosutinib 200 mg/day versus bosutinib 400/200 mg/day; Test type: Superiority or Other; p = 0.1234, Mixed Models Analysis; Median Difference (Final Values) = 1.83, 95% CI 2-sided [-0.50 to 4.22]
Statistical Analysis 3: Comparison: Bosutinib 200 mg/Day vs Placebo; Statistical Analysis 3 is comparison of annualized rate of kidney enlargement: placebo versus bosutinib 200 mg/day; Test type: Superiority or Other; p = 0.0050, Mixed Models Analysis; Median Difference (Final Values) = 3.06, 95% CI 2-sided [0.93 to 5.23]
Statistical Analysis 4: Comparison: Bosutinib 400 mg/Day vs Placebo; Statistical Analysis 4 is comparison of annualized rate of kidney enlargement: placebo versus bosutinib 400 mg/day; Test type: Superiority or Other; p = 0.1336, Mixed Models Analysis; Median Difference (Final Values) = 3.41, 95% CI 2-sided [-1.03 to 8.05]
Statistical Analysis 5: Comparison: Bosutinib 400/200 mg/Day vs Placebo; Statistical Analysis 5 is comparison of annualized rate of kidney enlargement: placebo versus bosutinib 400/200 mg/day; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Median Difference (Final Values) = 4.95, 95% CI 2-sided [2.65 to 7.30]

2. Secondary Outcome: Change From Baseline in Estimated Glomerular Filtration Rate (eGFR) at Months 12, 24, 25 and Early Termination
Description: eGFR was centrally evaluated. Glomerular filtration rate (GFR) is an index of kidney function that describes the flow of filtered fluid through the kidney. The Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation was used to calculate eGFR. Month 25 is the end of the ITPV.
Time Frame: Baseline, Month 12, Month 24, Month 25 (end of ITPV), and early termination
Population: The mITT population included all participants who were randomized and received at least 2 weeks' worth of treatment and have at least 1 post-randomization follow-up MRI assessment; n=the number of participants analyzed at that time point in the respective arms.
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Bosutinib 200 mg/Day | Bosutinib 400 mg/Day | Bosutinib 400/200 mg/Day | Placebo
Number analyzed (Participants) | 58 | 31 | 24 | 56
mL/min/1.73m^2
  CFB at Month 12 (n=26,4,21,31) | -6.38 (11.60) | -7.56 (11.27) | -11.52 (10.86) | 1.30 (9.71)
  CFB at Month 24 (n=23,3,20,30) | -8.47 (15.02) | -21.59 (13.74) | -13.16 (13.41) | -7.95 (12.91)
  CFB at End of ITPV (n=23,3,20,30) | -5.00 (10.78) | -13.24 (12.45) | -9.92 (14.55) | -2.74 (18.01)
  CFB at Early Termination (n=6,3,1,4) | -11.91 (8.79) | 0.78 (4.83) | -10.24 (NA) — Standard deviation (SD) was not calculated as only 1 participant was analyzed. | -2.75 (21.35)

3. Secondary Outcome: Time to First Occurrence or Worsening of Hypertension
Description: The time to first occurrence or worsening of hypertension was observed (defined as the need for increased dose of or need for additional anti-hypertensive medication). The numbers presented correspond to the very first occurrence or worsening of hypertension in that treatment group.
Time Frame: Baseline up to Month 25 (end of ITPV)
Population: The mITT-2 population included all participants who were randomized and received at least 2 weeks' worth of treatment and have at least 1 post-randomization follow-up MRI assessment (elimination of 1-month washout requirement).
Measure: Number; unit: days
Arm/Group | Bosutinib 200 mg/Day | Bosutinib 400 mg/Day | Bosutinib 400/200 mg/Day | Placebo
Number analyzed (Participants) | 58 | 31 | 24 | 56
days | 15 | 180 | 90 | 30

4. Secondary Outcome: Time to First Occurrence or Worsening of Back and/or Flank Pain
Description: The time to first occurrence or worsening of back and/or flank pain was observed (defined as initial onset of polycystic kidney disease [PKD]-related chronic back and/or flank pain; initiation of pain medication treatment for PKD-related chronic back and/or flank pain; addition of a pain medicine for treatment of PKD-related chronic back and/or flank pain; increase in dose of pain medication for treatment of PKD-related chronic back and/or flank pain). The numbers presented correspond to the very first occurrence or worsening of back and/or flank pain in that treatment group.
Time Frame: Baseline up to Month 25 (end of ITPV)
Population: as for outcome 3
Measure: Number; unit: days
Arm/Group | Bosutinib 200 mg/Day | Bosutinib 400 mg/Day | Bosutinib 400/200 mg/Day | Placebo
Number analyzed (Participants) | 58 | 31 | 24 | 56
days | 30 | 30 | 270 | 15

5. Secondary Outcome: Time to First Occurrence of Gross Hematuria
Description: Gross hematuria is the presence of blood in the urine (defined as pink, red, or cola-colored urine due to the presence of red blood cells). The numbers presented correspond to the very first occurrence of gross hematuria in that treatment group.
Time Frame: Baseline up to Month 25 (end of ITPV)
Population: as for outcome 3
Measure: Number; unit: days
Arm/Group | Bosutinib 200 mg/Day | Bosutinib 400 mg/Day | Bosutinib 400/200 mg/Day | Placebo
Number analyzed (Participants) | 58 | 31 | 24 | 56
days | 330 | 180 | 180 | 45

6. Secondary Outcome: Time to First Occurrence of Proteinuria
Description: Proteinuria is the presence of an excess of serum proteins in the urine, which may be an early sign of kidney disease. The numbers presented correspond to the very first occurrence of proteinuria in that treatment group.
Time Frame: Baseline up to Month 25 (end of ITPV)
Population: as for outcome 3
Measure: Number; unit: days
Arm/Group | Bosutinib 200 mg/Day | Bosutinib 400 mg/Day | Bosutinib 400/200 mg/Day | Placebo
Number analyzed (Participants) | 58 | 31 | 24 | 56
days | 360 | NA — No proteinuria events were observed. | 270 | 540

7. Secondary Outcome: Time to First Occurrence of End-Stage Renal Disease (ESRD) Requiring Dialysis >=56 Days
Description: ESRD is when the kidneys permanently fail to work at a level needed for daily life. No participants developed ESRD during the treatment period, therefore the analysis of the onset of ESRD requiring ≥56 days of dialysis was not performed.
Time Frame: Baseline up to Month 25 (end of ITPV)
Population: as for outcome 3
Measure: Number; unit: days
Arm/Group | Bosutinib 200 mg/Day | Bosutinib 400 mg/Day | Bosutinib 400/200 mg/Day | Placebo
Number analyzed (Participants) | 58 | 31 | 24 | 56
days | NA — No participants developed ESRD during the treatment period, therefore the analysis of the onset of ESRD requiring ≥56 days of dialysis was not performed. | NA — No participants developed ESRD during the treatment period, therefore the analysis of the onset of ESRD requiring ≥56 days of dialysis was not performed. | NA — No participants developed ESRD during the treatment period, therefore the analysis of the onset of ESRD requiring ≥56 days of dialysis was not performed. | NA — No participants developed ESRD during the treatment period, therefore the analysis of the onset of ESRD requiring ≥56 days of dialysis was not performed.

8. Secondary Outcome: Number of Participants With High Blood Urea Nitrogen (BUN) Levels
Description: A BUN test can reveal how well the kidneys are working by measuring the amount of urea nitrogen in the blood. A high BUN level (>1.3 times the upper limit of normal) may suggest that the kidneys are not working properly. Month 25 is the end of the ITPV.
Time Frame: Day 15, Months 6, 12, 18, 24, and 25 (end of ITPV)
Population: The safety analysis population included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Bosutinib 200 mg/Day | Bosutinib 400 mg/Day | Bosutinib 400/200 mg/Day | Placebo
Number analyzed (Participants) | 58 | 31 | 24 | 56
participants
  Day 15 | 0 | 0 | 2 | 0
  Month 6 | 0 | 0 | 0 | 0
  Month 12 | 0 | 0 | 0 | 0
  Month 18 | 0 | 0 | 0 | 0
  Month 24 | 0 | 0 | 1 | 0
  End of ITPV | 0 | 0 | 2 | 0

9. Secondary Outcome: Number of Participants With High Serum Creatinine (SCr) Levels
Description: A SCr test can reveal how well the kidneys are working by measuring the amount of urea nitrogen in the blood. A high SCr level (>1.3 times the upper limit of normal) may suggest that the kidneys are not working properly. Month 25 is the end of the ITPV.
Time Frame: Day 15, Months 6, 12, 18, 24, and 25 (end of ITPV)
Population: The safety analysis population included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Bosutinib 200 mg/Day | Bosutinib 400 mg/Day | Bosutinib 400/200 mg/Day | Placebo
Number analyzed (Participants) | 58 | 31 | 24 | 56
participants
  Day 15 | 0 | 1 | 0 | 0
  Month 6 | 0 | 0 | 0 | 0
  Month 12 | 0 | 0 | 0 | 1
  Month 18 | 0 | 0 | 0 | 0
  Month 24 | 0 | 1 | 1 | 1
  End of ITPV | 0 | 0 | 0 | 1

10. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Bosutinib
Time Frame: Day 1 (pre-dose and 1, 3, 5 and 24 hours post-dose), Day 15 (pre-dose and 1, 2, 3, 4, 6, 8 and 24 hours post-dose)
Population: The pharmacokinetic (PK) parameter analysis population included all participants randomized and treated who had at least 1 of the PK parameters of primary interest; n=the number of participants analyzed at that time point in the respective arms.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Bosutinib 200 mg/Day | Bosutinib 400 mg/Day | Bosutinib 400/200 mg/Day
Number analyzed (Participants) | 58 | 31 | 24
nanograms per milliliter (ng/mL)
  Day 1 (n=58,31,24) | 32.61 (53) | 74.87 (47) | 84.57 (56)
  Day 15 (n=58,16,22) | 68.72 (43) | 127.90 (28) | 155.00 (31)

11. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Bosutinib
Time Frame: Day 1 (pre-dose and 1, 3, 5 and 24 hours post-dose), Day 15 (pre-dose and 1, 2, 3, 4, 6, 8 and 24 hours post-dose)
Population: The PK parameter analysis population included all participants randomized and treated who had at least 1 of the PK parameters of primary interest; n=the number of participants analyzed at that time point in the respective arms.
Measure: Median (Full Range); unit: hours
Arm/Group | Bosutinib 200 mg/Day | Bosutinib 400 mg/Day | Bosutinib 400/200 mg/Day
Number analyzed (Participants) | 58 | 31 | 24
hours
  Day 1 (n=58,31,24) | 3.00 [1.00 to 24.00] | 3.00 [2.80 to 23.80] | 4.86 [1.00 to 5.25]
  Day 15 (n=58,16,22) | 3.95 [0.00 to 25.60] | 3.00 [1.00 to 8.00] | 5.00 [1.00 to 8.12]

12. Secondary Outcome: Area Under the Concentration-Time Profile From Time 0 to the Dosing Interval (AUCtau) of Bosutinib
Description: Area under the concentration-time profile from time 0 to time tau, the dosing interval, where tau=24 hours.
Time Frame: Day 1 (pre-dose and 1, 3, 5 and 24 hours post-dose), Day 15 (pre-dose and 1, 2, 3, 4, 6, 8 and 24 hours post-dose)
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Bosutinib 200 mg/Day | Bosutinib 400 mg/Day | Bosutinib 400/200 mg/Day
Number analyzed (Participants) | 58 | 31 | 24
ng*hr/mL
  Day 1 (n=58,30,24) | 437 (48) | 1040 (49) | 1149 (50)
  Day 15 (n=58,16,22) | 1059 (45) | 2052 (36) | 2384 (34)

13. Secondary Outcome: Lowest Concentration Observed During the Dosing Interval (Cmin) of Bosutinib
Time Frame: Day 15 (pre-dose and 1, 2, 3, 4, 6, 8 and 24 hours post-dose)
Population: The PK parameter analysis population included all participants randomized and treated who had at least 1 of the PK parameters of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Bosutinib 200 mg/Day | Bosutinib 400 mg/Day | Bosutinib 400/200 mg/Day
Number analyzed (Participants) | 58 | 16 | 22
ng/mL | 25.15 (49) | 19.60 (20880) | 50.67 (50)

14. Secondary Outcome: Apparent Oral Clearance (CL/F) of Bosutinib
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time Frame: Day 15 (pre-dose and 1, 2, 3, 4, 6, 8 and 24 hours post-dose)
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Bosutinib 200 mg/Day | Bosutinib 400 mg/Day | Bosutinib 400/200 mg/Day
Number analyzed (Participants) | 58 | 16 | 22
L/hr | 188.8 (45) | 195.0 (36) | 167.8 (34)

15. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of Bosutinib
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Time Frame: Day 1 (pre-dose and 1, 3, 5 and 24 hours post-dose), Day 15 (pre-dose and 1, 2, 3, 4, 6, 8 and 24 hours post-dose)
Population: The PK parameter analysis population included all participants randomized and treated who had at least 1 of the PK parameters of primary interest. There was no sufficient data to well-characterize the terminal phase, therefore Vz/F was not reported.
Arm/Group | Bosutinib 200 mg/Day | Bosutinib 400 mg/Day | Bosutinib 400/200 mg/Day
Number analyzed (Participants) | 0 | 0 | 0

16. Secondary Outcome: Terminal Elimination Half-Life (t1/2) of Bosutinib
Description: t1/2 is the time measured for the plasma concentration to decrease by one half.
Time Frame: Day 1 (pre-dose and 1, 3, 5 and 24 hours post-dose), Day 15 (pre-dose and 1, 2, 3, 4, 6, 8 and 24 hours post-dose)
Population: The PK parameter analysis population included all participants randomized and treated who had at least 1 of the PK parameters of primary interest. There was no sufficient data to well-characterize the terminal phase, therefore t1/2 was not reported.
Arm/Group | Bosutinib 200 mg/Day | Bosutinib 400 mg/Day | Bosutinib 400/200 mg/Day
Number analyzed (Participants) | 0 | 0 | 0

17. Secondary Outcome: Observed Accumulation Ratio (Rac) of Bosutinib
Description: Observed accumulation ratio (Rac) was calculated as AUC from time 0 to 24 hours (Day 15) divided by AUC from time 0 to 24 hours (Day 1).
Time Frame: Day 15 (pre-dose and 1, 2, 3, 4, 6, 8 and 24 hours post-dose)
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Bosutinib 200 mg/Day | Bosutinib 400 mg/Day | Bosutinib 400/200 mg/Day
Number analyzed (Participants) | 58 | 16 | 22
ratio | 2.452 (36) | 2.280 (42) | 2.075 (41)

18. Secondary Outcome: Change From Baseline in Kidney Disease Quality of Life (KDQoL)-36 Scale Scores at Month 25
Description: The KDQoL-36 is a 36-item questionnaire on kidney disease-specific measure of patient-reported quality of life with 5 subscales: physical and mental functioning (items 1-12); burden of kidney disease subscale (items 13-16); symptoms and problems (items 17-28); effects of kidney disease on daily life subscale (items 29-36). The raw scores are transformed linearly to a range of 0 to 100, with higher scores indicating better quality of life.
Time Frame: Baseline and end of ITPV (Month 25)
Population: The mITT-2 population included all participants who were randomized and received at least 2 weeks' worth of treatment and have at least 1 post-randomization follow-up MRI assessment (elimination of 1-month washout); n=the number of participants analyzed in the respective arms.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bosutinib 200 mg/Day | Bosutinib 400 mg/Day | Bosutinib 400/200 mg/Day | Placebo
Number analyzed (Participants) | 42 | 9 | 24 | 43
units on a scale
  Burden of Disease: Baseline (n=42,9,24,43) | 84.23 (18.48) | 84.722 (20.99) | 79.43 (24.97) | 74.86 (30.21)
  Burden of Disease: CFB Month 25 (n=32,3,22,34) | -2.54 (15.70) | -2.08 (9.55) | 0.57 (15.90) | 1.84 (19.13)
  Kidney Disease Effects: Baseline (n=42,9,24,43) | 93.30 (8.58) | 92.01 (11.06) | 91.54 (11.53) | 90.41 (14.10)
  Kidney Disease Effects: CFB Month 25; n=32,3,22,34 | 1.07 (5.48) | 3.13 (5.41) | -0.57 (9.72) | 3.22 (9.50)
  SF-12 Mental Health: Baseline (n=42,9,24,43) | 54.31 (6.39) | 51.11 (12.87) | 50.19 (9.28) | 51.33 (8.58)
  SF-12 Mental Health: CFB Month 25 (n=32,3,22,34) | -1.50 (5.87) | 6.55 (6.30) | 1.34 (7.35) | 0.12 (10.25)
  SF-12 Physical Health: Baseline (n=42,9,24,43) | 50.52 (6.93) | 51.78 (6.40) | 49.64 (8.35) | 47.17 (10.93)
  SF-12 Physical Health: CFB Month 25 (n=32,3,22,34) | -0.28 (5.81) | -7.59 (7.63) | -2.33 (8.16) | 2.32 (8.34)
  Symptoms/Problems: Baseline (n=42,9,24,43) | 93.13 (6.96) | 93.69 (7.35) | 90.72 (9.31) | 90.86 (9.29)
  Symptoms/Problems: CFB Month 25 (n=32,3,22,34) | -2.42 (7.21) | -8.33 (9.19) | -3.75 (8.04) | 0.27 (9.31)

19. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 30 days after last dose that were absent before treatment or that worsened relative to pre-treatment state. AEs included both SAEs and non-SAEs.
Time Frame: Baseline up to 30 days after last study drug administration
Population: The safety analysis population included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Bosutinib 200 mg/Day | Bosutinib 400 mg/Day | Bosutinib 400/200 mg/Day | Placebo
Number analyzed (Participants) | 58 | 31 | 24 | 56
participants
  AEs | 56 | 30 | 23 | 51
  SAEs | 12 | 4 | 6 | 5

20. Other Pre Specified Outcome: Number of Participants With Laboratory Abnormalities Meeting the Criteria for Potential Clinical Concern
Description: The following laboratory parameters were analyzed: hematology (hemoglobin, hematocrit, red blood cell [RBC] count, RBC morphology, platelet count, white blood cell [WBC] count, total neutrophils, eosinophils, monocytes, basophils, lymphocytes); blood chemistry (blood urea nitrogen [BUN], creatinine, glucose, calcium, sodium, potassium, chloride, total bicarbonate, aspartate aminotransferase [AST], alanine aminotransferase [ALT], total bilirubin, alkaline phosphatase, uric acid, albumin, and total protein; urinalysis (pH, glucose, protein, blood, ketones, nitrites, leukocyte esterase, microscopy [if urine dipstick was positive for blood, protein, nitrites or leukocyte esterase]); others (coagulation panel, circulating immune complex, and complement activation).
Time Frame: Baseline up to 30 days after last study drug administration
Population: The safety analysis population included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Bosutinib 200 mg/Day | Bosutinib 400 mg/Day | Bosutinib 400/200 mg/Day | Placebo
Number analyzed (Participants) | 58 | 31 | 24 | 56
participants | 53 | 20 | 23 | 43

21. Other Pre Specified Outcome: Number of Participants With Potentially Clinically Significant Vital Signs Findings
Description: Vital signs assessment included pulse rate and blood pressure. Criteria for vital sign values meeting potential clinical concern included: supine/sitting pulse rate <40 or >120 beats per minute (bpm), standing pulse rate <40 or >140 bpm; systolic blood pressure (SBP) of >=30 millimeters of mercury (mm Hg) change from baseline in same posture or SBP <90 mm Hg, diastolic blood pressure (DBP) >=20 mmHg change from baseline in same posture or DBP <50 mm Hg.
Time Frame: Baseline up to 30 days after last study drug administration
Population: The safety analysis population included all participants who received at least 1 dose of study drug; n=the number of participants analyzed in the respective arms.
Measure: Number; unit: participants
Arm/Group | Bosutinib 200 mg/Day | Bosutinib 400 mg/Day | Bosutinib 400/200 mg/Day | Placebo
Number analyzed (Participants) | 58 | 31 | 24 | 56
participants
  Supine SBP <90 mm Hg (n=2,2,1,4) | 0 | 0 | 0 | 0
  Sitting SBP <90 mm Hg (n=58,29,24,54) | 0 | 0 | 1 | 0
  Supine DBP <50 mm Hg (n=2,2,1,4) | 0 | 0 | 0 | 0
  Sitting DBP <50 mm Hg (n=58,29,24,54) | 0 | 1 | 1 | 0
  Supine Pulse Rate <40 or >120 bpm(n=2,2,1,4) | 0 | 0 | 0 | 0
  Sitting Pulse Rate <40 or >120 bpm (n=58,29,24,54) | 1 | 0 | 0 | 0
  Supine SBP ≥30 mm Hg Decrease (n=2,2,1,4) | 0 | 0 | 1 | 0
  Sitting SBP ≥30 mm Hg Decrease (n=58,29,24,54) | 2 | 1 | 2 | 2
  Supine DBP ≥20 mm Hg Decrease (n=2,2,1,4) | 0 | 0 | 1 | 0
  Sitting DBP ≥20 mm Hg Decrease (n=58,29,24,54) | 12 | 3 | 3 | 5
  Supine SBP ≥30 mm Hg Increase (n=2,2,1,4) | 0 | 0 | 0 | 0
  Sitting SBP ≥30 mm Hg Increase (n=58,29,24,54) | 3 | 1 | 3 | 3
  Supine DBP ≥20 mm Hg Increase (n=2,2,1,4) | 0 | 0 | 0 | 0
  Sitting DBP ≥20 mm Hg Increase (n=58,29,24,54) | 5 | 3 | 5 | 5

22. Other Pre Specified Outcome: Number of Participants With Potentially Clinically Significant Electrocardiogram (ECG) Findings
Description: ECGs were centrally evaluated. ECG parameters included PR interval, QRS interval, and corrected QT interval using Fridericia's formula (QTcF). Criteria for ECG changes meeting potential clinical concern included: PR interval greater than or equal to (≥)300 milliseconds (msec) or ≥25% increase when baseline is greater than (>)200 msec and ≥50% increase when baseline is less than or equal to (≤)200 msec; QRS interval ≥200 msec or ≥25%/50% increase from baseline; and QTcF ≥450 msec or ≥30 msec increase.
Time Frame: Baseline up to 30 days after last study drug administration
Population: as for outcome 21
Measure: Number; unit: participants
Arm/Group | Bosutinib 200 mg/Day | Bosutinib 400 mg/Day | Bosutinib 400/200 mg/Day | Placebo
Number analyzed (Participants) | 58 | 31 | 24 | 56
participants
  PR Interval ≥300 msec (n=58,31,24,56) | 0 | 0 | 0 | 0
  QRS Complex ≥200 msec (n=58,31,24,56) | 0 | 0 | 0 | 0
  QTcF Interval 450-<480 msec (n=58,31,24,56) | 3 | 2 | 0 | 6
  QTcF Interval 480-<500 msec (n=58,31,24,56) | 0 | 0 | 0 | 0
  QTcF Interval ≥500 msec (n=58,31,24,56) | 0 | 0 | 0 | 0
  PR Interval ≥25/50% Increase (n=57,28,23,52) | 0 | 0 | 0 | 0
  QRS Complex ≥25/50% Increase (n=57,28,23,52) | 0 | 0 | 0 | 0
  QTcF Interval 30-<60 msec Increase (n=57,28,23,52) | 4 | 1 | 1 | 5
  QTcF Interval ≥60 msec Increase (n=57,28,23,52) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 30 days after last study drug administration
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Arm/Group | Bosutinib 200 mg/Day | Bosutinib 400 mg/Day | Bosutinib 400/200 mg/Day | Placebo
Serious Adverse Events (participants affected / at risk) | 12/58 | 4/31 | 6/24 | 5/56
Other Adverse Events (participants affected / at risk) | 56/58 | 30/31 | 23/24 | 50/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Bosutinib 200 mg/Day (N=58) | Bosutinib 400 mg/Day (N=31) | Bosutinib 400/200 mg/Day (N=24) | Placebo (N=56)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Peptic ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Subileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hepatitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0
Hepatitis C (Infections and infestations) | 1 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 1 | 0
Renal cyst infection (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 2 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 1 | 0 | 0
Amylase increased (Investigations) | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 1 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Intracranial aneurysm (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0
Psychosomatic disease (Psychiatric disorders) | 1 | 0 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal cyst haemorrhage (Renal and urinary disorders) | 1 | 1 | 1 | 0
Renal cyst ruptured (Renal and urinary disorders) | 0 | 1 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal haemorrhage (Renal and urinary disorders) | 1 | 0 | 0 | 0
Cervix disorder (Reproductive system and breast disorders) | 0/28 | 0/14 | 1/15 | 0/35
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Bosutinib 200 mg/Day (N=58) | Bosutinib 400 mg/Day (N=31) | Bosutinib 400/200 mg/Day (N=24) | Placebo (N=56)
Anaemia (Blood and lymphatic system disorders) | 7 | 4 | 5 | 2
Eosinophilia (Blood and lymphatic system disorders) | 3 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 2 | 1 | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 3 | 2 | 2 | 3
Abdominal pain (Gastrointestinal disorders) | 4 | 8 | 2 | 7
Abdominal pain upper (Gastrointestinal disorders) | 5 | 7 | 8 | 5
Constipation (Gastrointestinal disorders) | 2 | 2 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 26 | 26 | 18 | 11
Dyspepsia (Gastrointestinal disorders) | 6 | 2 | 3 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 3
Nausea (Gastrointestinal disorders) | 21 | 15 | 13 | 9
Vomiting (Gastrointestinal disorders) | 6 | 11 | 9 | 4
Asthenia (General disorders) | 1 | 1 | 3 | 1
Chest pain (General disorders) | 1 | 2 | 0 | 0
Fatigue (General disorders) | 4 | 8 | 2 | 6
Influenza-like illness (General disorders) | 2 | 1 | 3 | 6
Oedema peripheral (General disorders) | 2 | 1 | 1 | 3
Pain (General disorders) | 1 | 0 | 0 | 3
Pyrexia (General disorders) | 2 | 3 | 2 | 1
Hepatocellular injury (Hepatobiliary disorders) | 3 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 2 | 1 | 0 | 3
Bronchitis (Infections and infestations) | 3 | 2 | 2 | 3
Cystitis (Infections and infestations) | 0 | 0 | 3 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 3
Influenza (Infections and infestations) | 2 | 0 | 1 | 3
Nasopharyngitis (Infections and infestations) | 12 | 3 | 8 | 8
Pharyngitis (Infections and infestations) | 0 | 0 | 3 | 4
Rhinitis (Infections and infestations) | 2 | 0 | 2 | 2
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 6 | 4 | 7 | 7
Urinary tract infection (Infections and infestations) | 8 | 2 | 2 | 8
Vaginal infection (Infections and infestations) | 1/28 | 0/14 | 0/15 | 3/35
Viral infection (Infections and infestations) | 2 | 0 | 1 | 3
Vulvovaginal mycotic infection (Infections and infestations) | 1/28 | 0/14 | 1/15 | 1/35
Excoriation (Injury, poisoning and procedural complications) | 3 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 18 | 16 | 12 | 4
Amylase increased (Investigations) | 2 | 4 | 3 | 1
Aspartate aminotransferase increased (Investigations) | 17 | 11 | 6 | 3
Blood creatine phosphokinase increased (Investigations) | 11 | 3 | 6 | 5
Blood creatinine increased (Investigations) | 2 | 1 | 2 | 2
Blood lactate dehydrogenase increased (Investigations) | 0 | 2 | 0 | 0
Blood phosphorus decreased (Investigations) | 0 | 2 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 4 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 2 | 0
Lipase increased (Investigations) | 5 | 6 | 6 | 3
Weight increased (Investigations) | 0 | 2 | 3 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 4 | 4 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 0 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 0 | 1 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 2 | 1 | 8
Flank pain (Musculoskeletal and connective tissue disorders) | 10 | 5 | 0 | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 2 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 3
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/28 | 0/14 | 1/15 | 0/35
Dizziness (Nervous system disorders) | 7 | 2 | 4 | 3
Dysgeusia (Nervous system disorders) | 0 | 2 | 0 | 0
Headache (Nervous system disorders) | 9 | 3 | 2 | 12
Insomnia (Psychiatric disorders) | 3 | 1 | 0 | 1
Haematuria (Renal and urinary disorders) | 4 | 3 | 1 | 4
Proteinuria (Renal and urinary disorders) | 1 | 0 | 2 | 3
Renal failure acute (Renal and urinary disorders) | 2 | 1 | 2 | 0
Amenorrhoea (Reproductive system and breast disorders) | 0/28 | 0/14 | 1/15 | 0/35
Cervical dysplasia (Reproductive system and breast disorders) | 0/28 | 0/14 | 1/15 | 0/35
Menorrhagia (Reproductive system and breast disorders) | 1/28 | 0/14 | 1/15 | 1/35
Metrorrhagia (Reproductive system and breast disorders) | 1/28 | 0/14 | 1/15 | 0/35
Ovarian cyst (Reproductive system and breast disorders) | 0/28 | 1/14 | 0/15 | 1/35
Vaginal inflammation (Reproductive system and breast disorders) | 0/28 | 0/14 | 1/15 | 1/35
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 3 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 1 | 2
Acne (Skin and subcutaneous tissue disorders) | 4 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 1 | 3 | 3
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Hypertension (Vascular disorders) | 8 | 3 | 5 | 9
Hypotension (Vascular disorders) | 1 | 0 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.